CLINICAL TRIAL: NCT04634890
Title: Bialystok Exercise Study in Diabetes
Acronym: BESD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Medical University of Bialystok (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R-I- 002/469/2014
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes; PreDiabetes; Overweight; Obesity; Dyslipidemias
Keywords: exercise intervention; type 2 diabetes prevention; type 2 diabetes treatment; prediabetes; behavioural intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Overweight; Obesity; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Type 2 Diabetes (Other): Subjects with type 2 diabetes, diagnosed within the last 3-5 years, treated with metformin only as an anti-diabetic drug
  Interventions: Behavioral: Exercise intervention
- Prediabetes (Other): Subjects with prediabetes, defined as impaired fasting glucose or/and impaired glucose tolerance
  Interventions: Behavioral: Exercise intervention
- Normoglycemia (Other): Subjects with normal fasting glucose and normal glucose tolerance
  Interventions: Behavioral: Exercise intervention

INTERVENTIONS:
Behavioral: Exercise intervention — Supervised exercise intervention composed of mixed aerobic and strength activities, with the frequency of 3 sessions per week for 12 weeks, for a total number of trainings of 36.

SUMMARY:
The "Bialystok Exercise Study in Diabetes" (BESD), is an exercise intervention study, conducted by the Department of Endocrinology, Diabetology and Internal Medicine and Clinical Research Centre of the Medical University of Bialystok. In the project, sedentary males at different stages of dysglycemia living in the city of Bialystok participate in three months of an exercise intervention consisting of supervised training sessions at a local fitness centre. The aim of the study is to assess the effectiveness of the exercise intervention in patients at different stages of dysglycemia progression, including type 2 diabetes and prediabetes and compare the response between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age: 35-65 years old
* BMI: 25-35 kg/m2
* Male gender
* Ability of performing exercise trainings
* Sedentary lifestyle

Exclusion Criteria:

* Smoking
* Drug or alcohol addiction
* Any chronic disease (exceptions: hypertension, obesity with BMI ≤ 35 kg/m2, type 2 diabetes)
* Any chronic medications (exceptions: angiotensin-converting-enzyme inhibitors for hypertension and metformin in type 2 diabetics)
* Highly active lifestyle
* Medical contraindications to participate in planned exercise sessions

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-08-11 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Three months
  Haemoglobin A1c measured by the high-performance liquid chromatography (HPLC) method
Fasting glucose | Three months
  Fasting glucose concentration measured in plasma using the colorimetric method
2-hour glucose | Three months
  Glucose concentration at 2-hour of the oral glucose tolerance test, measured in plasma using the colorimetric method
Fasting insulin | Three months
  Fasting insulin concentration measured in plasma using the immunoradiometric assay (IRMA)
Lean body mass | Three months
  Total lean body mass measured using the whole-body dual-energy X-ray absorptiometry (DXA)
Fat mass | Three months
  Total body fat mass measured using the whole-body dual-energy X-ray absorptiometry (DXA)
Visceral Adipose Tissue mass | Three months
  Visceral adipose tissue mass measured using the whole-body dual-energy X-ray absorptiometry (DXA)
Weight | Three months
  Total body weight measured using standardized scale
HOMA-IR | Three months
  Homeostatic model assessment for insulin resistance
HOMA-beta | Three months
  Homeostatic model assessment of beta cell function
VO2max | Three months
  Maximal oxygen consumption measured during cardio-pulmonary exercise test on treadmill
Triglycerides (TG) | Three months
  Serum triglycerides concentration measured using colorimetric method
High-density lipoprotein cholesterol (HDL) | Three months
  Serum high-density lipoprotein cholesterol (HDL) concentration measured using colorimetric method
Low-density lipoprotein cholesterol (LDL) | Three months
  Serum low-density lipoprotein cholesterol (LDL) concentration measured using colorimetric method
Total cholesterol | Three months
  Serum total cholesterol concentration measured using colorimetric method

SECONDARY OUTCOMES:
Plasma metabolome | Three months
  Changes in plasma metabolites concentrations measured using untargeted metabolomics
Skeletal muscle metabolome | Three months
  Changes in skeletal muscle metabolites concentrations measured using untargeted metabolomics
Subcutaneous adipose tissue metabolome | Three months
  Changes in subcutaneous adipose tissue metabolites concentrations measured using untargeted metabolomics
Skeletal muscle transcriptome | Three months
  Changes in skeletal muscle gene and smallRNA expressions measured using untargeted transcriptomics
Subcutaneous adipose tissue transcriptome | Three months
  Changes in subcutaneous adipose tissue gene and smallRNA expressions measured using untargeted transcriptomics

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Centre, Medical University of Bialystok, Bialystok, Podlaskie Voivodeship, Poland